CLINICAL TRIAL: NCT01685580
Title: Evaluation of Non-Invasive Ventilation Preoperative Lung Resection Surgery
Brief Title: Non-Invasive Ventilation Preoperative Lung Resection Surgery
Acronym: préOVNI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RB 11.095 préOVNI
Record Dates: First submitted 2012-09-12; First posted 2012-09-14 (Estimated); Last update posted 2025-12-03 (Actual); Status verified 2018-09

CONDITIONS: Surgery for Primary Lung Cancer
Keywords: primary lung cancer; lobectomy; pneumonectomy; non-invasive ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Manufacturer VPAP ST (Experimental): 7 days minimum non-invasive ventilation at 2 levels of pressure (BPAP) to the intervention.
  Interventions: Device: Manufacturer (VPAP ST)
- No intervention (No Intervention): usual advice

INTERVENTIONS:
Device: Manufacturer (VPAP ST) — non-invasive ventilation in two pressure levels 7 days before surgery
  Arms: Manufacturer VPAP ST

SUMMARY:
Surgical treatment is the standard treatment for localized forms of lung cancer non-small cell. It allows a 5-year survival exceeding 50% for complete resection of the tumor. This is a heavy treatment, resulting in a mortality of 4 to 8% and a morbidity of 20-60%. Securing this procedure is a major public health issue. The non-invasive ventilation is a technique commonly used postoperatively in acute respiratory distress and in the treatment of sleep apnea syndromes. Through its effect on oxygenation and pulmonary function parameters, the non-invasive ventilation achieved during 7 days minimum before the intervention could significantly reduce postoperative complications in patients with an obstructive or restrictive disorder, obesity or chronic heart failure.

The aim of the study is to demonstrate that the non-invasive ventilation in two pressure levels achieved during at least 7 days before surgery lung resection (lobectomy or segmentectomy) halved the pulmonary and cardiovascular postoperative patients with obstructive ventilatory disorder or restrictive, obesity or chronic heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years, to benefit from surgery scheduled for lung resection (lobectomy or segmentectomy) for primary lung cancer and having signed an informed consent.

AND

* Trouble obstructive (FEV / FVC <70% and FEV <80% predicted)

Or restrictive (FVC <80% or TLC <80%)

Or decrease in the ratio TLCO / VA <60%

Or history of respiratory failure with hypercapnic Pa CO2> 45 mmHg in the year preceding surgery

Or long-term oxygen

Or heart failure (clinical signs of heart failure and LVEF <55% or disorder of relaxation on echocardiography or atrial fibrillation)

Or history of acute cardiogenic pulmonary edema.

Or obesity (BMI> 30 kg/m2)

Exclusion Criteria:

* Inability to consent
* Patient declared inoperable given the comorbidities or refusing surgery or with unresectable tumors.
* Patient operable but with no comorbidities described in the inclusion criteria
* Contraindications to the non-invasive ventilation:

  * Lack of understanding of the technical
  * facial malformation
  * Tight stenosis of the upper airway
  * uncontrollable vomiting
  * Unable to remove the mask
  * Cognitive impairment or severe psychiatric jeopardizing the observance of the NAV
* Patient non-insured
* Patient already on invasive ventilation or non-invasive
* During Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-10-08 (Actual); Primary Completion 2017-10-25 (Actual); Study Completion 2017-10-25 (Actual)

PRIMARY OUTCOMES:
Reduction of pulmonary complications and cardiovascular postoperative | 1 month
  Demonstrate that the non-invasive ventilation in two pressure levels achieved during at least 7 days before surgery lung resection (lobectomy or segmentectomy) halved the pulmonary and cardiovascular postoperative patients with obstructive ventilatory disorder or restrictive, obesity or chronic heart failure.

SECONDARY OUTCOMES:
Identifying sub-groups of patients | 1 month
  Identify subgroups of patients benefiting most from a non-invasive ventilation preoperatively and safety of this technique preoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas PALEIRON, MD, Principal Investigator — Brest, Inter Army Hospital Clermont-Tonnerre
Locations (15):
- France (15):
  - Centre Hospitalier du Pays d'Aix, Aix-en-Provence, France
  - Centre Hospitalier Victor Dupouy, Argenteuil, France
  - Clinqiue du Grand Large, Brest, France
  - Hôpital Pontchaillou, Rennes, France
  - CHU de Rouen, Rouen, France
  - Hôpital Nord Ouest Villefranche Sur Saône, Villefranche-sur-Saône, France
  - CHU Angers, Angers
  - CHRU de Brest - Hôpital Morvan, Brest
  - Inter Army Hospital, Clermont-Tonnerre, Brest
  - Inter Army Hospital, Clamart
  - CHI Créteil, Créteil
  - CHU Limoges, Limoges
  - Hospital, Pasteur, Nice
  - CHU Saint-Etienne, Saint-Etienne
  - Inter Army Hospital, Saint-Anne, Toulon

REFERENCES:
- [Result] Paleiron N, Grassin F, Lancelin C, Tromeur C, Margery J, Natale C, Couturaud F; GFPC Group. Assessment of preoperative noninvasive ventilation before lung cancer surgery: The preOVNI randomized controlled study. J Thorac Cardiovasc Surg. 2020 Oct;160(4):1050-1059.e3. doi: 10.1016/j.jtcvs.2019.09.193. Epub 2019 Nov 23. PMID 31924365